CLINICAL TRIAL: NCT02304211
Title: Intra-Arterial Microdosing: Proof-of-Concept in Humans
Acronym: IAM-POC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00056933
Record Dates: First submitted 2014-11-26; First posted 2014-12-01 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: Microdosing; Phase 0; Exploratory Investigational New Drug (IND); Intra-Arterial; PET Imaging
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intra-Arterial Microdose Insulin (Experimental): Healthy volunteers will receive microdose insulin intra-arterially into the radial artery.
  Interventions: Drug: Insulin
- Systemic Insulin (Active Comparator): Healthy volunteers will receive full-dose insulin intra-venously.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Insulin will be administered either into the radial artery (microdose intervention) or IV (systemic intervention).

SUMMARY:
The purpose of this protocol is to demonstrate that intra-arterial administration of a drug can generate information in a manner that faithfully mimics effects of systemic administration but with little or no systemic effects.

DETAILED DESCRIPTION:
IAM is a novel approach combining the methodologies and techniques of 'microdosing' and 'intra-arterial drug delivery' to test new drugs in targeted organs or tissues. The main feature of this approach is that when a microdose (defined as 1/100th of the total body minimal pharmacological dose) is given into a body area 1/100th of the total body mass - a temporary pharmacological concentration is generated in that area that may be sufficient to generate and detect a biomarker relevant to the drug's safety and efficacy. The drug then returns systemically and is diluted to become a subpharmacological microdose. The significance of the approach is in the ability to obtain information on novel drugs in humans in a safe manner.

Insulin will be administered into the radial artery and compared with systemic administration. The effects on the ipsilateral hand will be compared with systemic effects and effects on the contralateral hand. The outcomes will be insulin pharmacokinetics, glucose and potassium levels, and 18F fluorodeoxyglucose (FDG) uptake as measured with Positron Emission Tomography (PET) imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
2. Healthy, non-smoking male subjects, 18 - 40 years of age with a BMI of 18 - 32 kg/m2 [BMI is rounded to the nearest tenth - a BMI of 32.045 should be rounded up to 32.05, which also would be rounded up to 32.1 and subject would be excluded; a BMI of 32.044 should be rounded down to 32.04 which would also be rounded down to 32.0 and the subject would be included].
3. Subject's health status will be determined by the medical history, physical examination, vital signs, electrocardiogram, blood chemistry, hematology, and urinalysis performed at screening.
4. Subjects must be willing to fast a minimum of 8 hours.
5. Subjects must be willing to abstain from alcohol from 2 days prior to Day 1 of the study until discharge.
6. Subjects must be willing to remain in the clinical research unit for the inpatient portion of the study from admission to discharge on Day 1.
7. Subjects must agree not to donate blood, plasma, platelets, or any other blood components during the study and for 4 weeks after completion of the study.
8. Renal function (creatinine clearance [CLcr] > 80 mL/min as calculated using the Cockcroft-Gault equation using lean body weight [LBW]) (Cockcroft and Gault 1976)
9. Subjects must have adequate arterial and venous access for receiving intra-arterial insulin infusions and placement of intravenous catheters for the collection of biomarker samples; and a positive Allen Test.

Exclusion Criteria:

1. Subjects with laboratory results outside the normal range, if considered clinically significant by the Investigator.
2. Hemoglobin concentration < 12.0 g/dL.
3. A mental capacity that is limited to the extent that the subject cannot provide legal consent or understand information regarding the potential risks of the study procedures and potential side effects of the investigational product.
4. Currently abusing drugs or alcohol or with a history of drug or alcohol abuse within the past two years.
5. Unwillingness or lack of ability to comply with the protocol or cooperate fully with the Principal Investigator and site personnel.
6. Use of any of the following:

   1. Any concomitant medication. Subjects who have received any prescribed or non-prescribed (over-the-counter [OTC]) systemic, topical, or oral medications, herbal or vitamin supplements within 14 days from Day 1. St. John's Wort (hypericin) must not have been taken for at least 30 days prior Day 1.
   2. Any drugs, foods or substances known to interfere with the acute effects of insulin or the biomarkers being evaluated within 14 days prior to Day 1.
7. Caffeine-or xanthine-containing products for 24 hours prior to Day 1 until discharged.
8. Use of alcohol for 48 hours prior to Day 1 until discharged.
9. Clinically significant ECG abnormality in the opinion of the Investigator.
10. Vital signs or clinically significant laboratory values at the screening visit that in the opinion of the Investigator would make the subject an inappropriate candidate for the study.
11. Has taken any investigational drug during the previous 30 days (or 5 half-lives, whichever is longer) prior to the screening visit or is currently participating in another investigational clinical trial.
12. Made any significant (as assessed by the investigator) donation (including plasma) or have had a significant loss of blood within 90 days prior to Day 1.
13. History or manifestation of clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, pulmonary, metabolic, endocrine, hematologic or other medical disorders.
14. Serious mental or physical illness within the past year.
15. History of regular alcohol consumption within 6 months of the study defined as:

    a. An average weekly intake of >14 drinks. One drink is equivalent to 12 g of alcohol: 12 ounces (360mL) of beer, 5 ounces (150mL) of wine or 1.5 ounces (45mL) of 80 proof distilled spirits.
16. Failure to agree to abstain from alcohol from 2 days before dosing.
17. Positive results on tests for drugs of abuse, cotinine or alcohol (breathalyzer) at screening or the assessment at check-in on Day 1.
18. Subjects who have used tobacco products or nicotine-containing products (including smoking cessation aids, such as gums or patches) within 6 months prior consenting.
19. History of sensitivity to insulin, 18F-FDG or other drugs (lidocaine) or other significant allergy that, in the opinion of the physician, contraindicates participation. This includes sensitivity to heparin or heparin-induced thrombocytopenia, if heparin is be used to maintain catheter patency.
20. Subjects who, in the opinion of the Investigator, should not participate in the study.
21. Subjects who are employed by the DCRU
22. Subjects who have a history of unexplained syncope; i.e., autonomic dysfunction (vasovagal syncope) or from blood collections.
23. Subjects who have a history of symptomatic hypotension and symptomatic hypoglycemia from fasting.
24. Lack of ability to understand verbal and/ or written English
25. History of clinically significant illness within 4 weeks prior to Day 1
26. Receipt of a transfusion or any blood products within 90 days prior to Screening.
27. Has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Glucose Plasma Levels | 2 hours
18F-FDG Uptake as measured with Positron Emission Tomography (PET) imaging | 2 hours

SECONDARY OUTCOMES:
Potassium Plasma Levels | 2 hours
Lactic Acid Plasma Levels | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Noveck, M.D., Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
PET Imaging data presently being analyzed for presentation and final manuscript publication

REFERENCES:
- [Background] Burt T, Rouse DC, Lee K, Wu H, Layton AT, Hawk TC, Weitzel DH, Chin BB, Cohen-Wolkowiez M, Chow SC, Noveck RJ. Intraarterial Microdosing: A Novel Drug Development Approach, Proof-of-Concept PET Study in Rats. J Nucl Med. 2015 Nov;56(11):1793-9. doi: 10.2967/jnumed.115.160986. Epub 2015 Aug 27. PMID 26315828